CLINICAL TRIAL: NCT03426683
Title: Efficacy, Safety and Microbiota of Intestinal Microbiota Transplantation for Inflammatory Bowel Diseases
Brief Title: The Effect of Intestinal Microbiota Transplantation for Inflammatory Bowel Diseases
Acronym: IBD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhongshan Hospital Xiamen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017004
Record Dates: First submitted 2017-10-27; First posted 2018-02-08 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Inflammatory Bowel Disease(IBD)
Keywords: Inflammatory Bowel Disease(IBD); Ulcerative colitis(UC); Crohn's disease(CD); intestinal microbiota transplantation; microbiota
MeSH Terms: conditions — Inflammatory Bowel Diseases; Colitis, Ulcerative; Crohn Disease | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: an open label, parallel study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized IMT (Experimental): The patients will receive Standardized Intestinal Microbiota Transplantation(Standardized IMT). The IMT was given to mid-gut by nose-jejunum nutrition tube or capsules. It was given three times a week.
  Interventions: Other: Intestinal Microbiota Transplantation
- traditional drugs (No Intervention): The patients will receive traditional medicine treatment as usual.

INTERVENTIONS:
Other: Intestinal Microbiota Transplantation — the bacteria will be transplanted to mid-gut by nose-jejunum nutrition tube. Patients in this study will be assigned to receive standardized IMT three times or traditional medicine and would be followed up for at least 3 year.
  Arms: Standardized IMT

SUMMARY:
There are many limitations in the current treatments of Inflammatory Bowel Diseases(IBD) which includes Ulcerative Colitis（UC) and Crohn's Disease(CD). Some patients have no or little reaction to the traditional drugs. Now the investigators realized that the intestinal microbiota is closely associated with the development of Inflammatory Bowel Diseases. In recent years, a retrospective study showed that the overall efficiency of intestinal microbiota transplantation for IBD was 79%, the overall remission rate was 43%, which opened a new chapter in the treatment of IBD. So the standardized intestinal microbiota transplantation is considered to be simple but effective emerging therapies for the treatment of IBD. In this project the investigators intend to carry out a single-center, randomized, single-blind clinical intervention study. The investigators plan to recruit patients with IBD in China. The patients will be randomly divided into two groups, one group will be given treatment of standardized intestinal microbiota transplantation, the other will be simply treated with traditional drugs, followed up for at least 1 year. The investigators aim to determine the efficiency, durability and safety of Intestinal Microbiota Transplantation for IBD treatment, and further to explore which major bacteria may effect in this project.

DETAILED DESCRIPTION:
In this projects the investigators aim to re-establish a gut balance of intestinal microbiota through Standardized Intestinal Microbiota Transplantation for Ulcerative Colitis(UC) and Crohn's Disease(CD).Investigators have established a standardized isolation, store, and transport steps of fecal bacteria from donated fresh stool in the laboratory. Then the bacteria will be transplanted to mid-gut by nose-jejunum nutrition tube or capsules.Participants in this study will be assigned to receive Standardized Intestinal Microbiota Transplantation three times a week or traditional medicine and would be followed up for at least 1 year. The clinical symptoms, sign, blood tests, endoscopy and questionnaire will be used to assess the efficiency, durability and safety of Standardized Intestinal Microbiota Transplantation at the start and end of the projects. At last, investigators will use 16S-rDNA to estimate the change of intestinal microbiota.

ELIGIBILITY:
Inclusion Criteria:

* Standard or conventional medicine treatment ineffective of Inflammatory Bowel Diseases(IBD) patients
* IBD patients with recurrent symptoms
* IBD patients who had drug dependence or recurrence when reduced or discontinued use
* Untreated IBD patients who voluntarily received Standardized Intestinal Microbiota Transplantation(IMT)
* Written informed consent/assent as appropriate

Exclusion Criteria:

* IBD patients with contraindications for gastrointestinal endoscopy
* IBD patients with indication of surgery
* Moderate and severe renal injuty(serum creatinine>2mg/dL or 177mmol/L), moderate and severe chronic obstructive pulmonary disease, severe hypertension, cerebrovascular accident, congestive heart failure, unstable angina pectoris
* Other serious diseases that may interfere the recruitment or affect the survival, such as cancer or acquired immune deficiency syndrome
* Mentally or legally disabled person
* Preparing for pregnancy
* Medical or social condition which in the opinion of the principal investigator would interfere with or prevent regular follow up
* Participating in other clinical trials.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2017-11-21 (Actual); Primary Completion 2021-10-29 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
The change of the modified Mayo score | 1 month, 3 months, 6months, 12 months
  Clinical remission defined as modified Mayo score≦2. Change from baseline will be assessed at different timepoint.The endpoint of follow-up is the time of clinical recurrence.

SECONDARY OUTCOMES:
The change of CDAI | 1 month, 3 months, 6months,12 months
  Clinical remission defined as CDAI(Crohn's disease activity index )≦150.Change from baseline will be assessed at different timepoint. The endpoint of follow-up is the time of clinical recurrence.
Relief of gastrointestinal symptoms | 1 months, 3 months, 6 months, 12months
  The onset and duration of gastrointestinal symptoms will be assessed by "Evaluation Score Table of Gastrointestinal Symptoms".Change from baseline will be assessed at different timepoint.
Changes of gut microbiota | 1 months, 3 months, 6 months, 12months
  Alpha and Beta diversity of GI microbiota by High-throughput sequencing on baseline line and1 month, 3 months, 6months ,12 months after treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital Affiliated to Xiamen University, Xiamen, Fujian, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Q, Fan Y, Zhang B, Yan C, Zhang Q, Ke Y, Chen Z, Wang L, Shi H, Hu Y, Huang Q, Su J, Xie C, Zhang X, Zhou L, Ren J, Xu H. Capsulized Fecal Microbiota Transplantation Induces Remission in Patients with Ulcerative Colitis by Gut Microbial Colonization and Metabolite Regulation. Microbiol Spectr. 2023 Jun 15;11(3):e0415222. doi: 10.1128/spectrum.04152-22. Epub 2023 Apr 24. PMID 37093057
- [Derived] Chen Q, Fan Y, Zhang B, Yan C, Chen Z, Wang L, Hu Y, Huang Q, Su J, Ren J, Xu H. Specific fungi associated with response to capsulized fecal microbiota transplantation in patients with active ulcerative colitis. Front Cell Infect Microbiol. 2023 Jan 5;12:1086885. doi: 10.3389/fcimb.2022.1086885. eCollection 2022. PMID 36683707

DOCUMENTS (2):
  • Study Protocol (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT03426683/Prot_001.pdf
  • Informed Consent Form (2017-05-01): https://cdn.clinicaltrials.gov/large-docs/83/NCT03426683/ICF_000.pdf